CLINICAL TRIAL: NCT00078299
Title: Evaluation of the Age-Related Eye Disease Study (AREDS) Clinical Lens Grading System
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040128; 04-EI-0128
Record Dates: First submitted 2004-02-20; First posted 2004-02-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Cataract
Keywords: Cortical; Nuclear Sclerosis; Posterior Subcapsular; Photographic Methods; Reproducibility (intra and interobserver); Cataract; Agreement; Grading System
MeSH Terms: conditions — Cataract

SUMMARY:
This study will evaluate a system developed to grade the severity of age-related cataract, a common cause of vision loss in older adults. Cataract research requires methods to simply and accurately determine the type and severity of cataracts in order to develop new, possibly non-surgical, treatments.

Patients 50 years of age and older with one of the three major age-related cataract types (nuclear, cortical, and posterior subcapsular) may be eligible for this study. Participants will be recruited from among patients enrolled in other National Eye Institute protocols.

Participants will have their eyes examined independently by two ophthalmologists with a biomicroscope, a magnifying device routinely used during eye examinations. The doctors will use the new grading system to record if a cataract is present, and if so, how severe it is. The examination includes measurement of visual acuity (vision chart test) and examination of the lens, retina, pupils and eye movements. Photographs of the eye will be taken using a special camera that flashes a bright light in the eye.

DETAILED DESCRIPTION:
Standardized lens photography with centralized grading of photographs has been used in clinical trials and epidemiologic studies of cataract. While photographic grading systems have been shown to be reliable, they are too expensive and complex to use in many studies. For some large studies, especially those with many centers or those in which lens changes are of secondary concern, it would be useful to have a simple clinical lens grading system that is reliable and that can be used with minimal training of examiners. Several clinical lens grading systems have been developed and found to be reliable in the hands of dedicated lens researchers, but the systems have been difficult for other ophthalmologists to use reliably.

The Age-Related Eye Disease Study (AREDA) has developed a simplified clinical cataract grading system to assess the severity of nuclear, cortical and posterior subcapsular cataracts, the 3 main types of age-related cataract. The system is designed to require minimal examiner training for persons already proficient in the use of the slit lamp. A total 150 participants with cataracts of varying severity, who are already participating in other NEI protocols, will be recruited to evaluate the reliability of the system. After being dilated, each participant will have a lens grading performed independently by 2 examiners. To provide information on the validity of the clinical gradings, lens photographs will be taken and graded using the detailed AREDS system for grading photographs. The data will allow us to evaluate (1) the agreement between the AREDS clinical lens grading system and the AREDS photographic system of grading lens opacities, and (2) the agreement on assessment of cataract severity among opthalmologists (with varying subspecialty) using the AREDS clinical lens grading method.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient must understand and sign the informed consent.
2. Patient must be at least 18 years of age.
3. Pupillary dilation to at least 6 mm must be possible.
4. Patients must have at least one natural lens present.

EXCLUSION CRITERIA:

Patients below the age of 18 will be excluded from participation in this study of age-related cataract.

1. Any condition such as corneal opacification that precludes adequate slit lamp examination and photography of the lens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2004-02; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Steinberg EP, Javitt JC, Sharkey PD, Zuckerman A, Legro MW, Anderson GF, Bass EB, O'Day D. The content and cost of cataract surgery. Arch Ophthalmol. 1993 Aug;111(8):1041-9. doi: 10.1001/archopht.1993.01090080037016. PMID 8352686
- [Background] Age-Related Eye Disease Study Research Group. The age-related eye disease study (AREDS) system for classifying cataracts from photographs: AREDS report no. 4. Am J Ophthalmol. 2001 Feb;131(2):167-75. doi: 10.1016/s0002-9394(00)00732-7. PMID 11228291
- [Background] Chylack LT Jr, Leske MC, McCarthy D, Khu P, Kashiwagi T, Sperduto R. Lens opacities classification system II (LOCS II). Arch Ophthalmol. 1989 Jul;107(7):991-7. doi: 10.1001/archopht.1989.01070020053028. PMID 2751471